CLINICAL TRIAL: NCT03051087
Title: A Multicenter, Randomized, Treated-controlled, Parallel, Open Label Study to Compare and Evaluate the Efficacy and Safety of Ganilever PFS and Orgalutran® in Infertility Women for Assisted Reproductive Technologies
Brief Title: To Compare and Evaluate the Efficacy and Safety of Ganilever PFS(Prefilled Syringe) and Orgalutran®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-GNCL001
Record Dates: First submitted 2017-02-07; First posted 2017-02-13 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Controlled Ovarian Stimulation
MeSH Terms: interventions — ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ganilever (ganirelix acetate) (Experimental): Prefilled syringe / 0.25mg/0.5mL
  Interventions: Drug: Ganirelix acetate
- Orgalutran (ganirelix acetate) (Active Comparator): Prefilled syringe / 0.25mg/0.5mL
  Interventions: Drug: Ganirelix acetate

INTERVENTIONS:
Drug: Ganirelix acetate

SUMMARY:
to compare and evaluate the efficacy and safety of Ganilever PFS and Orgalutran® in infertility women for assisted reproductive technologies

ELIGIBILITY:
Inclusion Criteria:

* An adult female between the ages of 20 and 39 at the time of screening
* Patients whose mean menstrual cycle was between 25 and 35 days
* Patients whose FSH (follicle stimulating hormone) concentration does not exceed 13 mIU / mL at screening
* Patients diagnosed with infertility due to one or more of the following A. Trouble Factors B. Male Factors C. Unexplained D. Uterine factors
* Patients with previous IVF experience less than 3
* Patient who signed the written consent after hearing the explanation of the purpose, method and effect of the clinical trial

Exclusion Criteria:

* If the sperm donor (spouse or non-spouse) is a severe male factor (Non obstructive azoospermia)
* Patients who were diagnosed as PCOS (polycystic ovary syndrome) during screening
* Patient with abnormal uterine bleeding during screening
* Patients diagnosed with primary ovarian failure
* Patients who has ovarian cysts that are not related to PCOS during screening
* Patients with tubal hydrops
* Patients with untreated non-reproductive endocrine disease
* Patients with a deformity of the reproductive organs that can not be conceived, or fibroids of the uterus that can not be conceived (only for submucosal myoma)
* Patients with less than 2 ovaries (0 or1)
* Patients with ovarian, breast, uterus, hypothalamus, or pituitary malignancies
* Patients with BMI <18 or BMI> 30
* Patients with an LH concentration of less than 1.2mIU / mL during screening
* Poor ovarian responder by bologna criteria
* Patients with moderate or severe renal impairment (creatinine clearance <60 mL / min) or liver function impairment (ALT or AST,> 5 times normal)
* Patients who experienced Grade 4 or higher OHSS (ovarian hyperstimulation syndrome) before
* Patients who are contraindicated for pregnancy
* Patients being pregnant or lactating
* Patients with hypersensitivity to IP
* Patients who have participated in other medication-related clinical trials since enrollment in this study, or have participated in other clinical trials within 3 months (90 days) before enrolling in this trial

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | about 10 days after randomization

SECONDARY OUTCOMES:
Proportion of subjects with LH (luteinizing hormone) rise > 10 mIU/mL | about 8~9 days after randomization (visit 4)
Oocyte quality | Day of oocyte retrieval (about 10 days after randomization)
Total administration dosage (IU) of Follitrope® PFS | During 8~9 days after randomization (until administration hCG)
Total administration duration (day) of Follitrope® PFS | During 8~9 days after randomization (until administration hCG)
Total administration dosage (mL) of Ganilever PFS or Orgalutran® | From 4~5 days after randomization to 8~9 days after randomization
Total administration duration (day) of Ganilever PFS or Orgalutran® | From 4~5 days after randomization to 8~9 days after randomization
Fertilization rate (%) | Day of oocyte retrieval (about 10 days after randomization)
Implantation rate (%) | About 4~5 weeks after Embryo transfer
Chemical pregnancy (%) | About 2 weeks after oocyte retrieval
Clinical pregnancy (%) | About 4~5 weeks after Embryo transfer
Ongoing pregnancy (%) | About 10~11 weeks after oocyte retrieval

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - CHA Gangnam Medical Center, Seoul